CLINICAL TRIAL: NCT05159765
Title: Progressive Myopia Treatment Evaluation for NaturalVue Multifocal Contact Lens Trial
Acronym: PROTECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Visioneering Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTI-NVMF-MPC-RCT-001
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Placebo Comparator): Contact lens with refractive correction, single vision optic
  Interventions: Device: Single vision contact lenses
- Treatment (Experimental): Contact lens with refractive correction, multifocal optic
  Interventions: Device: Multifocal contact lenses

INTERVENTIONS:
Device: Single vision contact lenses — Wearing contact lenses during waking hours may alter the progression of myopia
  Arms: Control
Device: Multifocal contact lenses — Wearing contact lenses during waking hours may alter the progression of myopia
  Arms: Treatment

SUMMARY:
This is a multi-center, randomized, double-masked clinical trial. All study devices are market approved/cleared in the localities where the study is conducted. Subjects will be randomly assigned to wear NaturalVue Sphere single vision contact lenses (SVCL) or NaturalVue Multifocal (NVMF) soft contact lenses for a total of three years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 7 to <13 (inclusive) at the Screening/Baseline examination.
2. Meet the following refractive criteria determined by cycloplegic autorefraction at Screening/Baseline:

   * Spherical Equivalent Refractive Error (SERE): between -0.75 and -5.00 D inclusive.
   * Astigmatism: ≤ -0.75 D
   * Anisometropia: < 1.000

Exclusion Criteria:

1. Has previously worn or currently wears rigid or gas permeable contact lenses, including orthokeratology lenses,
2. Appears to exhibit poor personal hygiene, that, in the Investigator's opinion, might prevent safe contact lens wear.
3. Is currently, or within 30 days prior to this study has been, an active participant in another clinical study.
4. Current or prior use of bifocals, progressive addition lenses, atropine, pirenzepine, multifocal or specialized contact lenses, or ANY other myopia control treatment.
5. The Investigator for any reason considers that it is not in the best interest of the subject to participate in the study, including if the child is not mature enough to independently handle and care for soft contact lenses.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Refractive Error relative to Baseline | Baseline, 12, 24, 36 months
  Mean change in cycloplegic auto-refraction (D)

SECONDARY OUTCOMES:
Change in Axial Length | Baseline,12, 24, 36 months
  Mean change in Axial Length (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Tuan, OD, PhD, Study Chair — VTI
Locations (8):
- United States (4):
  - Fig Garden Optometry, Fresno, California
  - North Suburban Vision Consultants, Deerfield, Illinois
  - Cooper Eye Care, New York, New York
  - Bellaire Family Eye Care, Bellaire, Texas
- Canada (2):
  - Toronto Eye Care, Toronto, Ontario
  - University of Waterloo School of Optometry, Waterloo, Ontario
- Hong Kong Polytechnic University, Tsim Sha Tsui, Hong Kong
- Myopia Specialist Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No